CLINICAL TRIAL: NCT02150954
Title: A Randomized Comparison of Foley Bulb With Low Dose Pitocin Versus Foley Bulb With a Standard Incremental Infusion Protocol for the Induction of Labor
Brief Title: Foley Bulb With Low Dose Pitocin Versus Foley Bulb With a Standard Incremental Infusion Protocol for the Induction of Labor
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00001312
Record Dates: First submitted 2014-05-23; First posted 2014-05-30 (Estimated); Results first posted 2014-07-23 (Estimated); Last update posted 2023-10-26 (Actual); Status verified 2014-06

CONDITIONS: Induction of Labor
Keywords: induction of labor; pitocin; foley bulb
MeSH Terms: interventions — Oxytocin

ARMS (2):
- foley bulb induction with low dose pitocin (Active Comparator): Subjects in this arm will receive a standard infusion protocol of pitocin starting at 1 milliunit/minute (mius/min) and increasing 2 milliunits per minute every 30 minutes.
  Interventions: Drug: pitocin
- foley bulb with standard incremental pitocin infusion protocol (Active Comparator): Subjects in this arm will receive a fixed low dose pitocin infusion protocol of 2 mius/min.
  Interventions: Drug: pitocin

INTERVENTIONS:
Drug: pitocin
  Other Names: oxytocin

SUMMARY:
The purpose of this research study is to compare induction of labor using a foley catheter bulb with a low dose of oxytocin versus a foley catheter bulb with an increasing dose of oxytocin. A foley catheter bulb with or without oxytocin is a common method of labor induction in patients whose cervix is not significantly dilated or thinned out (effaced). Oxytocin (pitocin) is a medicine used to increase the number and strength of the womb's contractions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a singleton pregnancy
2. Term pregnancy (> 37 weeks gestation)
3. Age ≥ 18 years
4. Bishop score < 5
5. Contractions < 6/hr
6. Reassuring fetal heart tracing

Exclusion Criteria:

1. Rupture of membranes
2. Antepartum bleeding
3. Fetal death
4. Placenta previa or low lying placenta
5. Active genital herpes infection
6. Previous use of an induction or preinduction agent during the current pregnancy
7. EFW >4500 grams
8. Non reassuring fetal testing
9. Inability to pass foley through cervix
10. Prior cesarean section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chad Grotegut, MD, Principal Investigator — Duke University; Brennan Fitzpatrick, MD, Principal Investigator — Duke University

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 121 subjects enrolled. Of the 121 subjects 2 were screen failures and 2 subject were excluded after consent due to meeting exclusion criteria.
Groups:
- Foley Bulb Induction With Low Dose Pitocin: Subjects in this arm will receive a standard infusion protocol of pitocin starting at 1 milliunit/minute (mius/min) and increasing 2 milliunits per minute every 30 minutes.
  pitocin
- Foley Bulb With Standard Incremental Pitocin Infusion Protocol: Subjects in this arm will receive a fixed low dose pitocin infusion protocol of 2 mius/min.
  pitocin
Period: Overall Study
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Started | 58 | 59
Completed | 57 | 59
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol | Total
Number analyzed (Participants) | 57 | 59 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 59 | 116
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 59 | 116
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 32 | 61
  White | 13 | 14 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 12 | 25
Region of Enrollment [Number; unit: participants]
  United States | 57 | 59 | 116

OUTCOME MEASURES:

1. Primary Outcome: Time to the Second Stage of Labor
Description: The second stage of labor was defined as the time from complete cervical dilation to delivery of the fetus.
Time Frame: foley bulb placement until second stage of labor (during admission for delivery, up to approximately 4 days)
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
hours | 18.2 [13.6 to 27.8] | 14.6 [9.9 to 28.3]

2. Primary Outcome: Time to Delivery
Description: Time from foley balloon placement until neonate delivery
Time Frame: foley bulb placement until delivery (during admission for delivery, up to approximately 4 days)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
hours | 23.7 [13.8 to 30.1] | 19.1 [12.1 to 32.1]

3. Secondary Outcome: Rate of Cesarean Delivery
Description: Number of participants having a cesarean delivery
Time Frame: during admission for delivery, up to approximately 4 days
Measure: Number; unit: participants
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
participants | 22 | 20

4. Secondary Outcome: Time to Active Labor
Description: Active labor was defined as the presence of regular, painful contractions and a minimum of 2 cm cervical dilation and complete effacement in nulliparous women or a minimum of 4 cm cervical dilation in multiparous women.
Time Frame: during admission for delivery, up to approximately 4 days
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
hours | 9.3 [5.8 to 22.4] | 12.2 [6.7 to 23.1]

5. Secondary Outcome: Time to Foley Expulsion or Removal
Description: Time from foley balloon placement until the expulsion or removal of the foley balloon.
Time Frame: foley bulb placement until removal, up to 10 hours
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
hours | 4.5 [2.7 to 7.5] | 5.6 [3.3 to 8.8]

6. Secondary Outcome: Incidence of Uterine Hyperstimulation
Description: Uterine hyperstimulation (tachysystole) was defined as uterine contractions occurring greater than 12 in 20 minutes.
Time Frame: during admission for delivery, up to approximately 4 days
Measure: Number; unit: participants
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
participants | 7 | 11

7. Secondary Outcome: Neonatal Outcome: Birthweight
Time Frame: at time of birth (0 to 1 hour)
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
gram | 3065 (530) | 3180 (511)

8. Secondary Outcome: Neonatal Outcome: Placental Abruption
Description: number of participants with placental abruption
Time Frame: during admission for delivery, up to approximately 4 days
Measure: Number; unit: participants
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
participants | 0 | 0

9. Secondary Outcome: Neonatal Outcome: Late Fetal Heart Rate Decelerations
Description: Late fetal heart rate decelerations were defined as a gradual decrease in the fetal heart rate associated with uterine contraction with the nadir of the deceleration occurring after the peak of the contraction.
Time Frame: during admission for delivery, up to approximately 4 days
Measure: Number; unit: neonates
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Number analyzed (Participants) | 57 | 59
neonates | 14 | 8

ADVERSE EVENTS:
Arm/Group | Foley Bulb Induction With Low Dose Pitocin | Foley Bulb With Standard Incremental Pitocin Infusion Protocol
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/59
Other Adverse Events (participants affected / at risk) | 0/57 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes